CLINICAL TRIAL: NCT03866941
Title: Evaluation of Acute and Chronic Toxicity of Some Synthetic Cannabinoids in Assiut Psychiatric Hospitals (Clinical and Experimental Study)
Brief Title: Acute and Chronic Toxicity of Some Synthetic Cannabinoids in Assiut Psychiatric Hospitals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MKMAbdelrahim, assistant lecturer, Assiut University
Other Study IDs: syntheticcannabinoidsAssiut
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Epidemiologic Data of Some Synthetic Cannibinoids Toxicity in Patients Presenting at Assiut University Hospital, Psychiatric Hospital of Ministry of Health); Proportion of Acute and Chronic Abusers of Synthetic Cannibinoids Among Cases of Illicit Drugs Abuser in Studied Sites
Keywords: synthetic cannabinoids, Assiut, violence,acute,chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- synthetic cannibinoids users
  Interventions: Behavioral: causes of abuse synthetic cannibinoids

INTERVENTIONS:
Behavioral: causes of abuse synthetic cannibinoids — Epidemiological data (age, sex, residence, occupation, route of abuse, the cause of abuse and smoking) (2) Symptoms and signs (seizures, psychosis, hallucinations) (3) Injuries and their relation to violence (type of wound, type of instrument, number of injuries, external or internal injuries and assailant or victim).

SUMMARY:
Synthetic cannabinoids (SCs) are new human-made mind-altering chemicals which are similar to chemicals found in the marijuana plant; they are recent to be used recreationally, especially by young adults. This new generation of novel cannabinoid compounds have been developed to avoid drug control laws and routine cannabinoid blood tests

DETAILED DESCRIPTION:
Synthetic cannabinoids (SCs) are new human-made mind-altering chemicals which are similar to chemicals found in the marijuana plant; they are recent to be used recreationally, especially by young adults[1]. This new generation of novel cannabinoid compounds has been developed to avoid drug control laws and routine cannabinoid blood tests[2].

SCs are dissolved in ethanol or acetone and sprayed on plant material, which is then sold in packets as incense, herbal blends. These products are sold under a variety of names including "Spice," "K2," "Black Mamba," "Scooby Snax" and in Egypt is known as "Voodoo" and "Strox". The chemical constituents and concentrations of compounds vary between and within packages[3].

Voodoo is one of these synthetic Cannabinoids that newly emerged in Egypt targeting the youth causing many reported cases of toxicity. This made the Egyptian Ministry of Health in 2014 to list it in drug schedule 1 and warned traffickers and users that they are now under criminal penalties[4].

Hundreds of SC were categorized into many structural groups and can be detected by Gass chromatography such as adamantoylindoles, aminoalkylindoles, benzoylindoles, cyclohexylphenols, dibenzopyrans, naphthoylindoles, naphthylmethylindoles, naphthylmethylindenes, naphthoylpyrroles, phenylacetylindoles, tetramethylcyclopropyl ketone indoles, quinolinyl ester indoles, and indazole carboxamide compounds[5].

Usually, 0.5 to 3 g of finely cut green/brown plant material is presented in colorful and professionally designed packets. Various herbs such as Pedicularis densiflora, Nymphacea caerulea, Leonotis leonurus, Leonurus sibiricus, Carnavalia maritima, and Zornia latifolia were declared as ingredients [6].

Smoking is the most common reported route of administration of SCs, although oral, pulmonary (via vapourization) and rectal administration has been described[7].

SCs interact with CB1 and CB2 cannabinoid receptors and elicit cannabimimetic effects similar to Δ9-tetrahydrocannabinol (THC), the primary psychoactive constituent in cannabis[8]. Although SC drugs mimic the psychotropic effects of cannabis, their undesired effects are unpredictable and more severe than those associated with cannabis[9].

SCs can result in acute, chronic and withdrawal manifestations[10]. Similar to cannabis, the acute intoxication of SCs may induce manifestations such as relaxation, euphoria, perceptual alteration, altered sense of time, and mild cognitive impairments [11]. Other adverse effects include confusion, dizziness, drowsiness, agitation, irritability, nausea, vomiting, hallucinations, delusions, increased heart rate, hypertension, vertigo and mydriasis [12-14]. Less common cardiac effects include chest pain, myocardial infarction, cardiac arrest and acute kidney damage[15].

Cases of synthetic cannabis abuse were associated with the manifestation of violence in Egypt and worldwide [16, 17]. These cognitive alterations increase the risk of road accidents if cannabis or SC users drive while intoxication[18]. Moreover, Psychoactive substances are often regarded as possible contributing causal factors in cases of violent injuries, sexual abuse, and homicides[15].

ELIGIBILITY:
Inclusion Criteria:

1. All the cases with the primary diagnosis of acute or chronic synthetic cannabinoids toxicity will be included in the study.
2. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* 1- Patients with a history of any chronic disease (renal and hepatic). 2- Patients refuse to participate in the study. 3- Abuse to other drugs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all cases diagnosed as acute or chronic synthetic cannibinoids toxicity which admitted to Emergency unit, Neuro-PsychatryUniversity Hospital - Assiut University and Psychiatric hospital of ministry of health
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
proportion of acute and chronicsynthetic cannibinoids abuser among cases of illicit drugs abuser in studied sites. | 2 years
  the magnitude and spread of this new drug of abuse

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa Abdel Moneim, Study Director — assiut univesity
Locations (1):
- Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No